CLINICAL TRIAL: NCT02489240
Title: Efficacy Study of Vitamin D to Treat Contrast-induced Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Shi Yang, Shi Yang, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLAGH301
Record Dates: First submitted 2015-07-01; First posted 2015-07-02 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Contrast-induced Nephropathy
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D supplementation group (Experimental): drug: vitamin D3 tablets (Vigantoletten; Merck Pharma, Germany); the frequency: 2000 IU vitamin D3 tablets were taken daily; duration: study treatment was commenced 3 days before intervention and maintained for 3 days after the procedure.
  Interventions: Drug: vitamin D3 tablets
- Control group (Placebo Comparator): drug: placebo tablets; the frequency: 2000 IU placebo tablets were taken daily; duration: study treatment was commenced 3 days before intervention and maintained for 3 days after the procedure.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vitamin D3 tablets — 2000 IU vitamin D3 tablets were taken daily for 6 days
  Other Names: Vigantoletten
  Arms: Vitamin D supplementation group
Drug: placebo — 2000 IU placebo tablets were taken daily for 6 days
  Arms: Control group

SUMMARY:
The investigators planned to research the effect of vitamin D supplementation on the incidence of contrast-induced nephropathy in patients undergoing coronary angiography.

DETAILED DESCRIPTION:
Vitamin D is primarily generated in the skin, in response to direct absorption of ultraviolet B radiation. Vitamin D can also be obtained through fortified foods and oral supplements. Contrast-induced nephropathy (CIN) is a generally reversible form of acute kidney injury that occurs mostly within 2-3 days of exposure to contrast medium (CM). The estimated incidence of CIN ranges from 2%-50%, and coronary angiography (CAG) or percutaneous coronary intervention (PCI), or both, are associated with CIN in about half of cases. Recently low vitamin D status has been shown to be associated with increased risk of CIN. However, its effects on CIN patients remain unclear. The investigators planned to determine the efficacy of vitamin D on the incidence of contrast-induced nephropathy in patients undergoing coronary angiography. This study may shed light as to whether oral vitamin D supplementation can be an adjunct therapy in CIN patients.

ELIGIBILITY:
Inclusion Criteria:

* The main inclusion criteria were patients who underwent coronary angiography.

Exclusion Criteria:

* The exclusion criteria were as follows: patients with chronic renal failure, chronic liver disease, bone disorders, and/or thyroid disorders.
* Patients were also excluded if they were taking vitamin D3 tablets or other lipid-regulating drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
the prevalence of contrast-induced nephropathy | 48-72h after treatment
  The primary efficacy variable was the prevalence of CIN between the vitamin D group and the control group.

SECONDARY OUTCOMES:
a change in serum creatinine level | at 1, 2, 3 days after percutaneous coronary intervention
  The change in serum creatinine level was measured at 1, 2, 3 days after the procedure.

OTHER OUTCOMES:
differences in the incidences of treatment-emergent adverse events | 6 days after treatment
  Treatment-emergent adverse events (TEAEs): hypercalcemia, renal insufficiency, constipation

CONTACTS AND LOCATIONS:
Overall Officials: Yu Tang Wang, M.D., Study Chair — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Sahin I, Gungor B, Can MM, Avci II, Guler GB, Okuyan E, Biter H, Yildiz SS, Ayca B, Satilmis S, Dinckal MH. Lower blood vitamin D levels are associated with an increased incidence of contrast-induced nephropathy in patients undergoing coronary angiography. Can J Cardiol. 2014 Apr;30(4):428-33. doi: 10.1016/j.cjca.2013.12.029. Epub 2014 Jan 4. PMID 24680172
- [Result] Ari E, Kedrah AE, Alahdab Y, Bulut G, Eren Z, Baytekin O, Odabasi D. Antioxidant and renoprotective effects of paricalcitol on experimental contrast-induced nephropathy model. Br J Radiol. 2012 Aug;85(1016):1038-43. doi: 10.1259/bjr/16327485. PMID 22815410
- [Result] Sokol SI, Srinivas V, Crandall JP, Kim M, Tellides G, Lebastchi AH, Yu Y, Gupta AK, Alderman MH. The effects of vitamin D repletion on endothelial function and inflammation in patients with coronary artery disease. Vasc Med. 2012 Dec;17(6):394-404. doi: 10.1177/1358863X12466709. PMID 23184900